CLINICAL TRIAL: NCT05053243
Title: Clinical Validation of the AliveCor Kardia 12L and 6L Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13692
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Kardia 12L — The purpose of this study is to collect clinical validation data to support an FDA submission for a 510(k) for the Kardia 12L hardware which enables the simultaneous diagnostic quality recording of all 6 limb leads and any chest lead. We will be recording both Leads V2 and V4 in a sequential fashion along with the Limb leads and a simultaneous 12-lead ECG to validate the hardware and a Deep Neural Network model which expands the 7 leads into a complete 12-lead ECG. The 12-lead ECG used for validation of the recordings and the 12-lead synthesis model is the GE Cardiosoft System which is FDA cleared.

SUMMARY:
AliveCor (www.alivecor.com) has developed an ECG device (KardiaMobile) that interfaces with iOS and Android smartphones and tablets. This ECG consists of a lightweight hardware case with two metal electrodes that can snap onto the back of the phone and a software application. By holding the right finger(s) on the right electrode and the left finger(s) on the left electrode, an electrical circuit is completed and a lead-I, 30 second rhythm strip is created. KardiaMobile and a newer device, KardiaMobile 6L, were approved by FDA for ECG rhythm recording. Recently, AliveCor developed two new devices: Kardia 12L and Kardia 6L to record 12- lead and 6-lead ECGs, respectively. However, the data generated from the two new devices have not yet been validated for accuracy. The purpose of this study is to evaluate the accuracy of the ECGs recorded by AliveCor Kardia 12L and 6L devices. This will be compared to simultaneous standard of-care 12-lead ECG recordings. The ECGs will be analyzed for accuracy and statistical difference using root-mean-square error and cross correlation between the median beats.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 years old or older
2. Ability to sit for an ECG and AliveCor Kardia 12L and Kardia 6L recordings for 20 minutes

Exclusion Criteria:

1. Any internal stimulator that would generate electrical interference with the recording system of the AliveCor Kardia 12L or Kardia 6L.
2. Open chest wounds or recent (<30 days) surgery to the chest or abdomen.
3. Absence of any limb that would require modification of the lead set-up

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Agreement on QRS width between Kardia 12L and ECG | 30 seconds
  Quantitative analysis on QRS width will be performed on the median-beat ECGs derived from the recorded ECGs from both devices as well as 12-lead ECG for each study participant
Agreement on PR interval between Kardia 12L and ECG | 30 seconds
  Quantitative analysis on PR interval will be performed on the median-beat ECGs derived from the recorded ECGs from both devices as well as 12-lead ECG for each study participant
Agreement on QT interval between Kardia 12L and ECG | 30 seconds
  Quantitative analysis on QT interval will be performed on the median-beat ECGs derived from the recorded ECGs from both devices as well as 12-lead ECG for each study participant

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Stavrakis, MD, PhD, Study Director — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided